CLINICAL TRIAL: NCT01987869
Title: Relationship Between Elevated Serum Serotonin Levels in Symptomatic Patients With Hyperemezis
Brief Title: Hiperemezis and Serotonin Elevated Serum Serotonin Levels in Hyperemesis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2013-88
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Nausea; Vomiting; Markedly Reduced Food Intake; Severe Dehydration
Keywords: hiperemesis gravidarum,vomiting,serotonin levels,ketonuria
MeSH Terms: conditions — Nausea; Vomiting; Dehydration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Serotonin excretion was investigated in the nausea and vomiting associated with hiperemezis gravid arum.

DETAILED DESCRIPTION:
The occurrence of severe nausea and vomiting of early pregnancy (hiperemezis gravid arum) is estimated between 0.3% to 1% of all pregnancies. Although hiperemezis gravid arum has been recognized for a long time, its pathophysiologic mechanisms are still poorly understood. Many theories have been advocated, but to date none of these have been convincing.

It has been demonstrated that the nausea and vomiting associated with increased in serotonin liberation. This has provided a rationale for the treatment of these symptoms with specific serotonin antagonists.

The aim of this trial was to investigate the possible relationship between hiperemezis gravid arum and serotonin liberation.

ELIGIBILITY:
Inclusion Criteria:

* 6-14 week pregnant women
* nausea
* protracted vomiting
* inability to tolerate food intake accompanied by obvious dehydration
* severe enough to justify hospitalisation
* at least 2+ ketonuria on dipstick urinanalysis.

Exclusion Criteria:

* with metabolic disorders such as diabet, thyroid

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pregnant women between six and fourteen weeks
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-02 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
serum serotonin levels in hiperemezis gravidarum | 6-14week pregnancy

SECONDARY OUTCOMES:
ıs there any assosiation between serotonin levels and severity of symptoms in pregnant women with hiperemezis | 6-14week pregnancy

OTHER OUTCOMES:
ıs there any assosiation between other serum parameters includes estrogen,progesterone and serum beta hcg | 6-14week pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: hüseyin cengiz, md, Study Chair — Bakırkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakirkoy Dr Sadi Konuk Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)